CLINICAL TRIAL: NCT02790008
Title: Magnetic Resonance Imaging and Fibrosis: Histological and Functional Changes in Left Ventricular Function Caused by Aortic Valve Disease
Brief Title: Magnetic Resonance Imaging and Fibrosis
Acronym: MRF
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Eva Tamas, university lecturer, Linkoeping University
Other Study IDs: SLS-501331
Record Dates: First submitted 2016-04-26; First posted 2016-06-03 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Heart Valve Disease; Ventricular Function; Fibrosis
Keywords: echocardiography; magnetic resonance imaging; cardiopulmonary exercise test
MeSH Terms: conditions — Heart Valve Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endomyocardial biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic valve disease: Patients with aortic stenosis referred to surgery. Exclusion criteria are concomitant heart valve disease, congenital heart disease, hemodynamic instability, previous cardiac surgery, history of myocardial infarction and coronary artery disease.

SUMMARY:
Aortic valve disease causes impaired let ventricular function (LVF) due to hypertrophy, dilatation and diffuse myocardial fibrosis yet the prognostic effect of fibrosis, waiting time for operation and postoperative exercise training is presently unknown.

The investigators aim to (1) determine the changes in LVF for patients on the waiting list; (2) establish non-invasive diagnostics for diffuse myocardial fibrosis; (3) relate LVF to fibrosis and physical capacity.

The unique design (echocardiography, cardiopulmonary exercise test, cardiac magnetic resonance tomography and myocardial biopsy on the same patients) makes it possible to establish relationship between results of histology and imaging; quantifying and qualifying fibrosis in vivo, evaluate LVF vs. general cardiopulmonary function and optimize health care prior to and after operation.

DETAILED DESCRIPTION:
AORTIC VALVE DISEASE & VENTRICULAR FUNCTION Aortic valve disease is the most common valvular heart disease in Europe (46.4%). The valve can be stenotic (aortic stenosis, AS) or can leak (aortic regurgitation, AR). While mostly elderly patients suffer from AS (a steadily growing group due to the increasing population above 60 years), AR occurs in younger individuals (20-60 years in general) who are still working and have a long life expectancy. The current treatment is aortic valve replacement (AVR) and in Sweden approx. 1800 AVR are performed every year with an increasing tendency. AVR is a procedure with low mortality (1.7%) nevertheless there is limited information available about postoperative morbidity, physical performance and quality of life.

Present guidelines suggest surgery when patients are presented with symptoms and/or show impairment of LVF (increasing LV diameters, declining ejection fraction - EF). These are though fairly crude measures as both symptoms and LV dilatation occur late in the natural history of the disease. Furthermore, we found previously that symptoms and LVF did not correlate which warrants the quest for searching more precise indicators.

AS causes pressure and AR causes volume overload which the LV compensates by concentric or eccentric hypertrophy initially. As the disease progresses even histological changes present e.g. diffuse fibrosis. Regional fibrosis after myocardial infarction is known to cause impaired LVF. However, there is no information available in the medical literature on how diffuse myocardial fibrosis affects LVF and whether it would be reversible following prosthetic valve implantation.

Cardiac surgery always carries risks for complications (e.g. mortality, stroke, postoperative arrhythmias, infections etc.) and life with a prosthetic heart valve is not necessarily uncomplicated. Our previous studies showed that preoperative impairment of the LVF can be irreversible and, as Gjertson showed, can progress to heart failure despite operation. Postoperative heart failure has a profound impact on long-term prognosis.

FIBROSIS & CARDIAC MAGNETIC RESONANCE IMAGING (cMRI) Well defined ischemic scars visualized reliably on cMRI by late gadolinium enhancement making it a useful diagnostic modality for myocardial viability in the clinical practice. Currently, in-vivo information on diffuse myocardial fibrosis is limited and optimal imaging method for clinical use is not established yet.

BIOMARKERS Biomarkers of myocardial fibrosis and their use as diagnostic tool for heart failure have been emerging lately. However, their diagnostic or predictive value for diffuse myocardial fibrosis in AS patients is not studied yet. The present study examines diffuse myocardial fibrosis pre- and postoperatively in AS patients, thus providing possibility to evaluate if fibrosis biomarkers can contribute as diagnostic/predictive markers for diffuse myocardial fibrosis and/or myocardial remodeling.

Based on the hypothesis that amount and location of the fibrotic tissue can be connected to impairment of LVF in severe aortic valve disease. We aim to validate special sequences (developed in Linköping) of cardiac magnetic resonance imaging (cMRI) as a diagnostic tool and to get information about the reversibility of myocardial fibrosis.

In addition, we plan to survey the physical capacity by cardiopulmonary exercise testing (CPET) pre- and postoperatively and study the relationship between physical performance capacity, fibrosis and LVF.

METHODS During cMRI T1 and T2 mapping of three ventricular slices equally spaced in the short axis direction will be performed. Gadolinium contrast is given for renewed T1 mapping allowing the calculation of the distribution volume, which will be taken as a sign of fibrosis. Functional data are calculated from the cine images. Flow images are generated by 2D phase contrast recording of through-plane flow times the flow area produces an estimate of stroke volume and cardiac output. In a 4D phase contrast recording, LV inflow can be characterized in terms of four flow compartments as well as the presence or absence of vortices in the intraventricular flow pattern.

3D-QALAS (3D-quantification using an interleaved Look-Locker acquisition sequence with T2 preparation pulse) is based on a 3D spoiled Turbo Field Echo sequence using inversion recovery with interleaved T2 preparation. It allows rapid acquisition and provides quantitative information of both T1 and T2 relaxation times in the same scan with full coverage of the LV.

NT-proBNP, HsTnT, and markers for myocardial fibrosis are to be taken to assess relations between these parameters and fibrosis in the heart muscle.

Intraoperatively 5 biopsies (1.2 mm) are to be taken of the LV in a standardized fashion. Samples are to be dyed and analysed by an image quantification program for verification and quantification of fibrosis.

CPET records data about the cardiovascular and respiratory systems under stress simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* patients with aortic valve disease

Exclusion Criteria:

* concomitant cardiac co-morbidity,
* concomitant surgical intervention,
* symptomatic lung disease,
* mental or physical disability limiting participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 pts with severe AS but without any other concomitant heart valve disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Left ventricular function: | 1 year
  a composite measure of ejection fraction = EF (%); left ventricular wall thickness lateralt and septalt (mm), left ventricular volumes (ml)
Degree of fibrosis | 1 year
  semi-quantitative scale 1-4

SECONDARY OUTCOMES:
Diastolic Function | 1 year
  A composite measure of blood velocity through the mitral valve {E and A wave (cm/s) and E/A}, through the pulmonary veins in systole and diastole (cm/s) and tissue velocity in the lateral wall and the ventricular septum.
Physical capacity | 1 year
  Oxygen uptake measured by cardiopulmonary exercise test (ml/(kg x min)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Vascular and Cardiothoracic Surgery, University Hospital Linkoping, Linköping, Sweden

REFERENCES:
- [Derived] Nilsson H, Bellander C, Carlen A, Nylander E, Hedman K, Tamas E. Systolic blood pressure response during exercise testing in symptomatic severe aortic stenosis. Open Heart. 2025 Jan 21;12(1):e003084. doi: 10.1136/openhrt-2024-003084. PMID 39842940